CLINICAL TRIAL: NCT01691300
Title: C11-Acetate PET/CT in Multiple Myeloma: Added Value to F18-Fluorodeoxyglucose PET/CT for Staging and Response Assessment
Brief Title: C11-Acetate PET/CT in Multiple Myeloma: Added Value to F18-Fluorodeoxyglucose PET/CT
Acronym: ACTMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 99-2177A
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Myeloma
Keywords: C11-acetate PET/CT; Multiple myeloma; Pretreatment staging; Response assessment
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACT PET/CT (Experimental): Dual-tracer ACT/FDG PET/CT and WB-DCE-MRI at baseline (pretreatment), post-induction and post-ASCT (if eligible)
  Interventions: Other: ACT PET/CT

INTERVENTIONS:
Other: ACT PET/CT — Old tracer but new indication

SUMMARY:
Positron emission tomography combined with computed tomography using carbon-11 acetate (ACT PET/CT) may help detect lesions before treatment and evaluate response following therapy in patients with from multiple myeloma (MM). This study aimed to prospectively assess the clinical utility of ACT PET/CT in MM as compared to the commonly used F18-fluorodeoxyglucose(FDG).

ELIGIBILITY:
Inclusion Criteria:

* at least 20 years of age
* previously untreated
* complete pre-treatment clinical staging including bone marrow examination
* written informed consent to participate in the study

Exclusion Criteria:

* concurrent active malignant tumor(s)
* pregnant or breast feeding women
* non-compliant to PET/CT or to MRI
* marked renal impairment (contraindicated for contrast-enhanced MRI)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pretreatment lesion detection | Within 2 weeks before initiation of therapy
  Reference standards: bone marrow examination and whole-body dynamic contrast-enhanced MRI

SECONDARY OUTCOMES:
Post-induction response assessment | Approximately 4 months after initiation of therapy depending on the regimen
  Reference standard: clinical response based on International Uniform Criteria and bone marrow examination if any
Post-ASCT response assessment | Approximately 3 months after ASCT
  Reference standard: clinical response based on International Uniform Criteria and bone marrow examination if any

OTHER OUTCOMES:
Progression free survival | With 2 years of follow-up time
  Based on clinical follow-up (M-protein or FLC assay, bone marrow examination or imaging findings)

CONTACTS AND LOCATIONS:
Overall Officials: Chieh Lin, MD, PhD, Principal Investigator — Department of Molecular Imaging Center and Nuclear Medicine, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hostpial, Guishan, Taoyuan County, Taiwan